CLINICAL TRIAL: NCT05611151
Title: Real-time Computer-Aided Detection of Colonic Adenomas With NEC WISE VISION® Endoscopy: Prospective, Randomized Clinical Performance Evaluation
Brief Title: Real-time Computer-Aided Detection of Colonic Adenomas With NEC WISE VISION® Endoscopy
Acronym: COLOWISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NEC Corporation (Industry)
Collaborators: Meditrial Europe Ltd. (Industry); Meditrial USA Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: WV-2022-01
Record Dates: First submitted 2022-11-01; First posted 2022-11-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer; Adenoma Colon; Polyp of Colon
Keywords: Screening; Artificial Intelligence
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps

STUDY DESIGN:
Intervention Model Description: Parallel trial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- CADe Colonoscopy (Experimental): CADe Colonoscopy: Patient undergoes WISE VISION® Endoscopy CADe colonoscopy
  Interventions: Diagnostic Test: Computer Aided Detection (CADe)
- HDWL Colonoscopy (Active Comparator): HDWL Colonoscopy: Patient undergoes HDWL colonoscopy without CADe
  Interventions: Diagnostic Test: Computer Aided Detection (CADe)

INTERVENTIONS:
Diagnostic Test: Computer Aided Detection (CADe) — Computer-aided detection (CADe) devices are used in conjunction with colonoscopy to aid in the detection of lesions in the gastrointestinal tract.

SUMMARY:
This is a prospective, multicenter, randomized study to evaluate the clinical performance of a novel CADe device, WISE VISION® Endoscopy System, in patients undergoing high-definition white light (HDWL) colonoscopy for screening or surveillance of colorectal Cancer (CRC).

Eligible subjects who meet the study inclusion/exclusion criteria will be randomized in a 1:1 ratio to undergo colonoscopy :

* Experimental: CADe colonoscopy procedure with WISE VISION® Endoscopy (CADe Group)
* Control: Standard Colonoscopy without CADe (Standard Colonoscopy Group)

DETAILED DESCRIPTION:
This study aims to evaluate whether NEC WISE VISION® Endoscopy enhances the ability to detect mucosal lesions when compared with the current standard-of-care procedure (high-definition white light [HDWL] colonoscopy). The CADe device, Wise VISION® Endoscopy, contains an artificial intelligence/machine learning (AI/ML) advanced algorithm to aid the endoscopists in detection of colonic lesions.

This study plans to enrol 830 subjects aged ≥ 45 years and < 75 years, who are scheduled for screening or surveillance colonoscopy.

After review of the inclusion and exclusion criteria, eligible subjects will be randomized in a 1:1 ratio to receive either computer-aided colonoscopy (CADe Group) or standard colonoscopy without CADe (Standard Colonoscopy Group).

All adenomas, that are identified during the colonoscopies, will be removed and biopsied as per standard clinical practice to assess adenoma miss rate, polyp miss rate, adenomas per colonoscopy and other endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Patient is presenting to the endoscopy unit for colon cancer screening or surveillance colonoscopy.
* Signed Informed Consent

Exclusion Criteria:

1. Contraindications to colonoscopy
2. Colonoscopy within the previous three (3) years
3. High-risk indications for colonoscopy
4. Antithrombotic therapy that cannot be stopped, precluding polyp resection
5. Inflammatory bowel disease
6. Referred for endoscopic mucosal resection (EMR)
7. Familial adenomatous polyposis syndrome or Serrated Polyposis Syndrome
8. Pregnant or planning a pregnancy during the study period

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 830 (Actual)
Dates: Start 2023-04-30 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Adenomas per Colonoscopy (APC) | during the procedure/surgery
  Total number of histologically confirmed adenomas resected divided by the total number of colonoscopies.

CONTACTS AND LOCATIONS:
Overall Officials: Hitoshi Ikeda, Study Director — NEC Corporation
Locations (5):
- Kansas City VA Hospital, Kansas City, Missouri, United States
- GastroZentrum Lippe, Bad Salzuflen, Germany
- Italy (2):
  - Humanitas Mater Domini, Castellanza
  - Humanitas Research Hospital, Milan
- Portsmouth Hospitals University NHS Trust, Cosham, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yamada M, Saito Y, Imaoka H, Saiko M, Yamada S, Kondo H, Takamaru H, Sakamoto T, Sese J, Kuchiba A, Shibata T, Hamamoto R. Development of a real-time endoscopic image diagnosis support system using deep learning technology in colonoscopy. Sci Rep. 2019 Oct 8;9(1):14465. doi: 10.1038/s41598-019-50567-5. PMID 31594962
- See also: Meditrial Clinical Research Organization — http://meditrial.net